CLINICAL TRIAL: NCT01566292
Title: Intraprostatic Botulinum Toxin Type "A" Injection in Patients With Benign Prostatic Hyperplasia and Unsatisfactory Response to Medical Therapy: a Randomised, Double-blind, Controlled Trial Using Subjective and Objective Outcomes
Brief Title: Intraprostatic Botulinum Toxin Type "A" Injection in Patients With Benign Prostatic Hyperplasia and Unsatisfactory Response to Medical Therapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, PROFESSOR PIER FRANCESCO BASSI, Prof, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 268/08
Record Dates: First submitted 2012-03-09; First posted 2012-03-29 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Benign Prostatic Hyperplasia (BPH); Benign Prostatic Enlargement (BPE)
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BOTOX (Experimental)
  Interventions: Drug: BOTOX

INTERVENTIONS:
Drug: BOTOX — Botulinum Toxin type A, 200-300 UI dilued in 6 ml of saline solution
  Other Names: Botulinum toxin type A

SUMMARY:
The injection of botulinum neurotoxin A into the prostate represents an alternative, minimal invasive treatment in patient with lower urinary tract symptoms (LUTS) associated to benign prostatic hyperplasia (BPH).

Objective: To evaluate the effectiveness of BTA in treating patients with symptomatic BPH and unsatisfactory response to combined medical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Moderate-to-severe LUTS as determined by the International Prostate Symptom Score
* Mean peak urinary flow rate of no more than 15 mL/s with a voided volume of at least 150 mL, or postvoid residual urine volume (PVR) of more than 100 ml and urodynamic parameters indicative of bladder outlet obstruction (BOO) according to International Continence Society

Exclusion Criteria:

* Patients with neurogenic voiding disorders, prostate or bladder cancer, bladder stones, urethral stricture, chronic bladder catheterization were excluded from the study.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
evaluation of symptomatic improvement after treatment as measured by the IPSS score. A successful outcome was defined as a reduction of IPSS score of > 50% from baseline. | 3 month

SECONDARY OUTCOMES:
safety and tolerability of treatment | 3 month
  Quality of life improvement as measured by QoL score, changes in prostate volume, total PSA levels, maximal flow at uroflowmetry, post-void residual urine,maximal cystometric capacity, Bladder Outlet Obstruction Index, sexual modifications evaluated by International Index of Erectile Function.

CONTACTS AND LOCATIONS:
Overall Officials: PierFrancesco Bassi, Professor, Principal Investigator — Catholic University of sacred Heart
Locations (1):
- Catholic University of Sacred Heart, Rome, Italy

REFERENCES:
- [Result] Maria G, Brisinda G, Civello IM, Bentivoglio AR, Sganga G, Albanese A. Relief by botulinum toxin of voiding dysfunction due to benign prostatic hyperplasia: results of a randomized, placebo-controlled study. Urology. 2003 Aug;62(2):259-64; discussion 264-5. doi: 10.1016/s0090-4295(03)00477-1. PMID 12893330